CLINICAL TRIAL: NCT01871064
Title: Residual Curarization and Its Incidence at Tracheal Extubation in China
Acronym: RECITE-China
Status: Completed | Type: Observational
Sponsor: Xinmin Wu (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Xinmin Wu, Professor, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Other Study IDs: LCE50498
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Residual Curarization
Keywords: Laparotomy; laparoscopic surgery; general anesthesia; Neuromuscular Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: TOF-Watch SX® Monitoring of NMB — Participants will have the extent of NMB monitored by a TOF-Watch SX®.

SUMMARY:
This study will assess the residual neuromuscular blockade (NMB) Train-Of-Four (TOF) ratios at tracheal extubation when anesthesiologists have determined that full recovery of neuromuscular function has occurred using standard clinical criteria for participants whose non-depolarizing-induced NMB is either not reversed or reversed with an acetylcholinesterase inhibitor administered as per standard routine care.

DETAILED DESCRIPTION:
This is a prospective, multi-site, anesthesiologist and PACU nurse TOF-Watch SX® blinded observational study of surgical patients undergoing elective laparoscopic or open abdominal procedures requiring general anesthesia and non-depolarizing neuromuscular blockade. There are two temporal aspects to the data collection: a prospective data collection in the OR and PACU; and a retrospective chart review one week after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18;
* American Society of Anesthesiologists(ASA) class 1-3;
* Scheduled for elective open or laparoscopic abdominal surgery that is anticipated to last less than 4 hours;
* Administration of general anesthesia and ≥ 1 dose of non-depolarizing neuromuscular blockers for endotracheal intubation or maintenance of neuromuscular blockade;
* Planned for extubation to occur in the OR;
* Signed informed consent.

Exclusion Criteria:

* Redo surgery on the same hospital admission;
* Pre-established need or expected to require post-operative mechanical ventilation;
* Conditions, surgical procedures, or participant positioning that may interfere with TOF-Watch SX® operation, calibration, or accuracy;
* Anesthesiologist use of objective neuromuscular monitoring during surgery (e.g. mechanomyography, electromyography or related method);
* Pregnancy;
* Participation in any other clinical trial;
* Member or a family member of the personnel of the investigational or Sponsor staff directly involved with this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults 18 years of age or older scheduled to undergo an elective open abdominal or laparoscopic surgical procedure for an anticipated duration of less than four hours will be approached for participation in the study.
Sampling Method: Probability Sample
Enrollment: 1571 (Actual)
Dates: Start 2012-12; Primary Completion 2013-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Residual Neuromuscular Blockade (NMB)(Train of Four [TOF] Ratio <0.9) at Time of Tracheal Extubation | Immediately prior to tracheal extubation in the OR
  Neuromuscular functioning was monitored at time of tracheal extubation by applying three TOF electrical stimulations to the ulnar nerve and assessing twitch response at the adductor pollices muscle. T1 and T4 refer to the magnitudes (height) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0) indicates the extent of recovery from NMB, with a higher ratio indicating greater recovery from NMB. A T4/T1 Ratio of <0.9 is indicative of residual NMB.

SECONDARY OUTCOMES:
Percentage of Participants With Residual NMB (TOF Ratio <0.9) Upon Arrival to the Post-anesthesia Care Unit (PACU) | Immediately upon PACU arrival
  Neuromuscular functioning was monitored at time of PACU arrival by applying three TOF electrical stimulations to the ulnar nerve and assessing twitch response at the adductor pollices muscle. T1 and T4 refer to the magnitudes (height) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0) indicates the extent of recovery from NMB, with a higher ratio indicating greater recovery from NMB. A T4/T1 Ratio of <0.9 is indicative of residual NMB.
Percentage of Participants With Residual NMB at Various TOF Ratios (<0.6, ≥0.6 to <0.7, ≥0.7 to <0.8, ≥0.8 to <0.9) at Tracheal Extubation | Immediately prior to tracheal extubation in the OR
  Neuromuscular functioning was monitored at time of tracheal extubation by applying three TOF electrical stimulations to the ulnar nerve and assessing twitch response at the adductor pollices muscle. T1 and T4 refer to the magnitudes (height) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0) indicates the extent of recovery from NMB, with a higher ratio indicating greater recovery from NMB
Percentage of Participants With Residual NMB at Various TOF Ratios (<0.6, ≥ 0.6 to <0.7, ≥ 0.7 to <0.8, ≥0.8 to <0.9) Upon Arrival to the PACU | Immediately upon PACU Arrival
  Neuromuscular functioning was monitored at time of PACU arrival by applying three TOF electrical stimulations to the ulnar nerve and assessing twitch response at the adductor pollices muscle. T1 and T4 refer to the magnitudes (height) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0) indicates the extent of recovery from NMB, with a higher ratio indicating greater recovery from NMB.

CONTACTS AND LOCATIONS:
Overall Officials: Xinmin Wu, MD, Principal Investigator — Peking University First Hospital
Locations (32):
- China (32):
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - ZhuJiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College of HUST, Wuhan, Hubei
  - Wuhan Union Hospital, Wuhan, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Northern Jiangsu Province People's Hospital, Yangzhou, Jiangsu
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Xijing Hospital, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Xinjiang Traditional Chinese Medicine Hospital, Ürümqi, Xinjiang
  - First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Second Affiliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang
  - Peking University First Hospital, Beijing
  - Beijing Tongren Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Renji Hospital, Shanghai
  - Ruijin Hospital, Shanghai
  - Shanghai Cancer Hospital, China, Shanghai
  - Shanghai First People's Hospital, Shanghai
  - Shanghai Zhongshan Hospital, Shanghai

REFERENCES:
- [Background] Aldrete JA. The post-anesthesia recovery score revisited. J Clin Anesth. 1995 Feb;7(1):89-91. doi: 10.1016/0952-8180(94)00001-k. No abstract available. PMID 7772368
- [Background] Murphy GS, Szokol JW, Franklin M, Marymont JH, Avram MJ, Vender JS. Postanesthesia care unit recovery times and neuromuscular blocking drugs: a prospective study of orthopedic surgical patients randomized to receive pancuronium or rocuronium. Anesth Analg. 2004 Jan;98(1):193-200. doi: 10.1213/01.ANE.0000095040.36648.F7. PMID 14693617
- [Background] Apfel CC, Laara E, Koivuranta M, Greim CA, Roewer N. A simplified risk score for predicting postoperative nausea and vomiting: conclusions from cross-validations between two centers. Anesthesiology. 1999 Sep;91(3):693-700. doi: 10.1097/00000542-199909000-00022. PMID 10485781
- [Background] Murphy GS, Brull SJ. Residual neuromuscular block: lessons unlearned. Part I: definitions, incidence, and adverse physiologic effects of residual neuromuscular block. Anesth Analg. 2010 Jul;111(1):120-8. doi: 10.1213/ANE.0b013e3181da832d. Epub 2010 May 4. PMID 20442260
- [Background] Murphy GS, Szokol JW, Marymont JH, Franklin M, Avram MJ, Vender JS. Residual paralysis at the time of tracheal extubation. Anesth Analg. 2005 Jun;100(6):1840-1845. doi: 10.1213/01.ANE.0000151159.55655.CB. PMID 15920224
- [Background] Fezing AK, d'Hollander A, Boogaerts JG. Assessment of the postoperative residual curarisation using the train of four stimulation with acceleromyography. Acta Anaesthesiol Belg. 1999;50(2):83-6. PMID 10418647
- [Background] Debaene B, Plaud B, Dilly MP, Donati F. Residual paralysis in the PACU after a single intubating dose of nondepolarizing muscle relaxant with an intermediate duration of action. Anesthesiology. 2003 May;98(5):1042-8. doi: 10.1097/00000542-200305000-00004. PMID 12717123
- [Background] Kopman AF, Yee PS, Neuman GG. Relationship of the train-of-four fade ratio to clinical signs and symptoms of residual paralysis in awake volunteers. Anesthesiology. 1997 Apr;86(4):765-71. doi: 10.1097/00000542-199704000-00005. PMID 9105219
- [Background] Bissinger U, Schimek F, Lenz G. Postoperative residual paralysis and respiratory status: a comparative study of pancuronium and vecuronium. Physiol Res. 2000;49(4):455-62. PMID 11072806
- [Background] Sundman E, Witt H, Olsson R, Ekberg O, Kuylenstierna R, Eriksson LI. The incidence and mechanisms of pharyngeal and upper esophageal dysfunction in partially paralyzed humans: pharyngeal videoradiography and simultaneous manometry after atracurium. Anesthesiology. 2000 Apr;92(4):977-84. doi: 10.1097/00000542-200004000-00014. PMID 10754616
- [Background] Eriksson LI, Sundman E, Olsson R, Nilsson L, Witt H, Ekberg O, Kuylenstierna R. Functional assessment of the pharynx at rest and during swallowing in partially paralyzed humans: simultaneous videomanometry and mechanomyography of awake human volunteers. Anesthesiology. 1997 Nov;87(5):1035-43. doi: 10.1097/00000542-199711000-00005. PMID 9366453
- [Background] Royse CF, Newman S, Chung F, Stygall J, McKay RE, Boldt J, Servin FS, Hurtado I, Hannallah R, Yu B, Wilkinson DJ. Development and feasibility of a scale to assess postoperative recovery: the post-operative quality recovery scale. Anesthesiology. 2010 Oct;113(4):892-905. doi: 10.1097/ALN.0b013e3181d960a9. PMID 20601860
- [Background] Fuchs-Buder T, Claudius C, Skovgaard LT, Eriksson LI, Mirakhur RK, Viby-Mogensen J; 8th International Neuromuscular Meeting. Good clinical research practice in pharmacodynamic studies of neuromuscular blocking agents II: the Stockholm revision. Acta Anaesthesiol Scand. 2007 Aug;51(7):789-808. doi: 10.1111/j.1399-6576.2007.01352.x. PMID 17635389
- [Derived] Yu B, Ouyang B, Ge S, Luo Y, Li J, Ni D, Hu S, Xu H, Liu J, Min S, Li L, Ma Z, Xie K, Miao C, Wu X; RECITE-China Investigators. Incidence of postoperative residual neuromuscular blockade after general anesthesia: a prospective, multicenter, anesthetist-blind, observational study. Curr Med Res Opin. 2016;32(1):1-9. doi: 10.1185/03007995.2015.1103213. Epub 2015 Nov 11. PMID 26452561